CLINICAL TRIAL: NCT00573573
Title: Phase 1 Study to Evaluate the Efficacy of Using Energy Specific Far Infrared Radiation Treatment for Hyperparathyroidism.
Brief Title: Energy Specific Far Infrared Radiation Treatment for Hyperparathyroidism
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GAAD Medical Research Institute Inc. (Other)
Responsible Party: Dr. Kwasi Donyina/Founder and President, GAAD Medical Research Institute Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAAD-HT-CTP1
Record Dates: First submitted 2007-12-12; First posted 2007-12-14 (Estimated); Last update posted 2009-03-24 (Estimated); Status verified 2009-03

CONDITIONS: Hyperparathyroidism
Keywords: PRIMARY HYPERPARATHYROIDISM; PARATHYROID NEOPLASMS; SECONDARY HYPERPARATHYROIDISM; HYPOCALCEMIA
MeSH Terms: conditions — Hyperparathyroidism; Hyperparathyroidism, Primary; Parathyroid Neoplasms; Hyperparathyroidism, Secondary; Hypocalcemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Radiation: Far Infrared Radiation

INTERVENTIONS:
Radiation: Far Infrared Radiation — Far Infrared Radiation (5μm to 20μm wavelength) for 30 to 40 minutes each session.

SUMMARY:
A study to determine the possibility of using far infrared radiation to treat Hyperparathyroidism.

DETAILED DESCRIPTION:
Overactive parathyroid glands secrete an excess of parathyroid hormones, resulting in increased levels of calcium in the blood stream, which can lead to weakening of the bones and to kidney stones.

We are postulating that the non-invasive energy specific electromagnetic radiation of the central nervous system, the viscera and the endocrine system has the potential to stop the over secretion of the parathyroid hormones and normalize the body's metabolic functions.

ELIGIBILITY:
Inclusion Criteria:

* Persons with parathyroid disease

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-03 (Estimated); Study Completion 2009-07 (Estimated)

PRIMARY OUTCOMES:
The primary end point is to determine the therapeutic effects of far infrared radiation on Hyperparathyroidism. | 2 years

SECONDARY OUTCOMES:
Effect of far infrared radiation treatment on other immune deficiency diseases like thyroidism and diabetes | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ken Nedd, M.D., Study Director — GAAD Medical Research Institute Inc.; Kwasi Donyina, Ph.D., Study Chair — GAAD Medical Research Institute Inc.
Locations (1):
- The Centre for Incurable Diseases, Toronto, Ontario, Canada